CLINICAL TRIAL: NCT01444339
Title: Study of Two Investigational Pneumococcal Vaccines in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PPR05
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Pneumococcal Infections; Streptococcus Pneumoniae Infections; Pneumococcal Pneumonia
Keywords: Pneumococcal Infections; Streptococcus Pneumoniae Infections; Pneumococcal Vaccine
MeSH Terms: conditions — Pneumococcal Infections; Pneumonia, Pneumococcal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Pneumococcal Vaccine Formulation 1 (Experimental): Participants will receive an injection of pneumococcal vaccine (Formulation 1, 1 middle dose) on Day 0 and Day 30, respectively.
  Interventions: Biological: Pneumococcal Vaccine Formulation 1
- Pneumococcal Vaccine Formulation 2 (Experimental): Participants will receive an injection of Pneumococcal vaccine (Formulation 2, 2 low doses) on Day 0 and Day 30, respectively.
  Interventions: Biological: Pneumococcal Vaccine Formulation 2
- Pneumococcal Vaccine Formulation 3 (Experimental): Participants will receive an injection of pneumococcal vaccine (Formulation 3, 2 middle doses) on Day 0 and Day 30, respectively.
  Interventions: Biological: Pneumococcal Vaccine Formulation 3
- Pneumococcal Vaccine Formulation 4 (Experimental): Participants will receive an injection of pneumococcal vaccine (Formulation 4, 2 middle doses) on Day 0 and Day 30, respectively.
  Interventions: Biological: Pneumococcal Vaccine Formulation 4
- Pneumococcal Vaccine Formulation 5 (Experimental): Participants will receive an injection of pneumococcal vaccine (Formulation 5, 2 high doses) on Day 0 and Day 30, respectively.
  Interventions: Biological: Pneumococcal Vaccine Formulation 5
- Pooled placebo Group (Placebo Comparator): Participants will receive an injection of a placebo on Day 0 and Day 30, respectively.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Pneumococcal Vaccine Formulation 1 — 0.5 mL, intramuscular (1 middle dose)
  Arms: Pneumococcal Vaccine Formulation 1
Biological: Pneumococcal Vaccine Formulation 2 — 0.5 mL, intramuscular (2 low doses)
  Arms: Pneumococcal Vaccine Formulation 2
Biological: Pneumococcal Vaccine Formulation 3 — 0.5 mL, intramuscular (2 middle doses)
  Arms: Pneumococcal Vaccine Formulation 3
Biological: Pneumococcal Vaccine Formulation 4 — 0.5 mL, intramuscular (2 middle doses)
  Arms: Pneumococcal Vaccine Formulation 4
Biological: Pneumococcal Vaccine Formulation 5 — 0.5 mL, intramuscular (2 high doses)
  Arms: Pneumococcal Vaccine Formulation 5
Biological: Placebo — 0.5 mL, intramuscular
  Other Names: Tris buffered saline
  Arms: Pooled placebo Group

SUMMARY:
This study is designed to evaluate the safety, tolerability, and immunogenicity of two investigational pneumococcal vaccines at three dose levels in healthy adults.

Primary Objective:

- To evaluate the safety and tolerability of two investigational pneumococcal vaccines.

Observational Objective:

- To evaluate the immunogenicity of the investigational pneumococcal vaccines.

DETAILED DESCRIPTION:
An initial cohort of 6 participants will receive a single dose of one of two investigational pneumococcal vaccines. After safety evaluation of that cohort, additional cohorts will receive 2 injections 30 days apart of same investigational pneumococcal vaccine at same or increased dose level. All participants will be monitored for safety for 30 days after each vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 50 years on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and comply with all trial procedures
* Subject is healthy, as determined by medical history and physical examination
* For a woman of child-bearing potential, use of an effective method of contraception or abstinence from at least 4 weeks prior to first vaccination until 4 weeks after the last vaccination.

Exclusion Criteria:

* Known pregnancy or positive serum/urine pregnancy test
* Currently breastfeeding a child
* Chronic illness, that in the opinion of the investigator, is at a stage that could interfere with trial conduct or completion
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccine components or history of a life threatening reaction to the trial vaccine(s) or to a vaccine containing any of the same substances
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with the assessment of immune response
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination
* Planned receipt of any vaccine in the 4 weeks following the trial vaccination
* Known seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C
* Laboratory confirmed / self-reported thrombocytopenia contraindicating intramuscular vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Identified as a study site employee who is involved in the protocol and may have direct access to trial-related data
* Previous vaccination against pneumococcal disease (in the previous 5 years)
* History of pneumococcal infection (confirmed either clinically, serologically, or microbiologically) within 5 years
* At high risk for pneumococcal infection during the trial
* Living in a household with children < 5 years of age.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants reporting solicited injection site reactions, solicited systemic reactions, unsolicited systemic reactions, and serious adverse events occurring throughout the trial | 30 days post-vaccination
  Solicited injection site reactions: Pain, Erythema, and Swelling. Solicited systemic reactions: Fever (Temperature), Headache, Malaise, and Myalgia

SECONDARY OUTCOMES:
Immunogenicity of Investigational Pneumococcal vaccines after 2 vaccinations | Days 0 and 30 post-vaccination
  Evaluation of immune responses to antigen component of the investigational vaccine by enzyme linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Ltd.
Locations (1):
- Allschwil, Switzerland

REFERENCES:
- [Derived] Bologa M, Kamtchoua T, Hopfer R, Sheng X, Hicks B, Bixler G, Hou V, Pehlic V, Yuan T, Gurunathan S. Safety and immunogenicity of pneumococcal protein vaccine candidates: monovalent choline-binding protein A (PcpA) vaccine and bivalent PcpA-pneumococcal histidine triad protein D vaccine. Vaccine. 2012 Dec 14;30(52):7461-8. doi: 10.1016/j.vaccine.2012.10.076. Epub 2012 Nov 2. PMID 23123106
- See also: Related Info — http://www.sanofipasteur.com